CLINICAL TRIAL: NCT02759666
Title: A Multicenter, Open-Label, Phase 1 Trial of SHR3162 Given Orally to Subjects With Advanced Solid Tumors
Brief Title: A Phase I Trial of SHR3162 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR3162-002
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Neoplasm; Solid Tumors
Keywords: PARP; advanced solid tumor
MeSH Terms: conditions — Neoplasms | interventions — fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SHR3162 (Experimental): 3 to 6 participants (traditional "3+3" design) will be enrolled in 6 dose levels. SHR3162 was administered once daily in dose levels 1 and 2 and will be administered twice daily in dose levels 3 to 6.
  Interventions: Drug: SHR3162

INTERVENTIONS:
Drug: SHR3162 — SHR3162 capsule(s) is administered orally QD.
  Other Names: Fluzoparib

SUMMARY:
This is an open-label, multicenter, non-randomized, dose-escalation phase 1 trial to evaluate the safety and tolerability of SHR3162 in participants with advanced solid tumors.

DETAILED DESCRIPTION:
Poly adenosine diphosphate (ADP)-ribose polymerase (PARP) is a family of proteins that plays important roles in multiple cellular processes, including single-strand DNA breaks, which if left unrepaired, leads to double-strand breaks (DSB) during DNA replication. The DSB can be repaired either through error-free homologous recombination (HR) or error-prone non-homology end joining. In HR deficient cancer cells with mutations on HR genes such as BRCA1, BRCA2 or partner and localizer of BRCA2 (PALB2), DSB cannot be efficiently and correctly repaired, resulting in cell death. Viable cells, on the other hand, have normal HR and do not replicate as often as cancer cells; thus they can survive PARP inhibition. PARP inhibitors are being actively developed worldwide as promising anti-tumor therapeutics. The current trial will be conducted in participants with advanced solid tumors for whom satisfactory treatments are not yet available.

In the dose-escalation phase, patients will be enrolled sequentially into the 8 dose levels of SHR3162 designated in this study(3-6 patients per cohort). One to two sentinel participants in Cohort 1 who will be treated and closely monitored for 24 hours. If no adverse effects are noted during the 24-hour period, dosing of further participants in the cohort may continue.

In the dose expansion part of the study, up to 12 additional participants will be enrolled at the MTD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18.
2. Ability to understand the purposes and risks of the trial and his/her signed informed consent form approved by Human Research Ethics Committee (HREC) of the trial site was obtained before the entering the trial.
3. Histologically or cytologically confirmed advanced or metastatic solid tumor for which no established standard therapy is available.
4. At least one measurable lesion by CT or MRI according to RECIST Version 1.1, which is not in irradiated area (only for expansion phase).
5. Recovered from toxicities of prior anti-cancer treatment to Grade 1 or less (in case of alopecia, Grade 2 is acceptable).
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Life expectancy of at least 3 months.
8. Acceptable liver function defined below:

   * Total bilirubin ≤1.5 times upper limit of normal (ULN);
   * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 times ULN; however, ≤5 times ULN in a participant who has liver metastases or is treated with biliary drainage
9. Acceptable renal function defined below:

   * Serum creatinine ≤1.5 times ULN or calculated creatinine clearance (by the Cockcroft-Gault formula) ≥60 mL/minutes
10. Acceptable coagulation status defined below:

    * Prothrombin time <1.3 times ULN
    * Partial thrombin time <1.3 times ULN
11. Acceptable hematologic status (without hematologic supports including hematopoietic factor, blood transfusion) defined below:

    * Absolute neutrophil count (ANC) ≥1500/μL
    * Platelet count ≥100000/μL
    * Hemoglobin ≥9.0 g/dL
12. No clinically significant abnormalities in urinalysis.
13. Female participants of child bearing potential agree not to be pregnant or lactating during the study and for three months following the last dose of study drug. Both men and women of reproductive potential must agree to use a highly effective method of birth control during the study and for three months following the last dose of study drug. A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly.

Exclusion Criteria:

1. Hematologic malignancies.
2. Cardiac disease with New York Heart Association (NYHA) Class III or IV, including congestive heart failure, myocardial infarction within 6 months prior to the trial entry, unstable arrhythmia, or symptomatic peripheral arterial vascular disease.
3. Previously treated malignancies other than the current disease, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years at the trial entry.
4. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
5. Major surgery, other than diagnostic surgery, within 4 weeks prior to the trial entry, without complete recovery.
6. Percutaneous coronary intervention conducted within 6 months prior to the trial entry for cardiac infarction or angina pectoris.
7. Seizure disorders requiring anticonvulsant therapy.
8. Taking a medication that prolongs QT interval and has a risk of Torsade de Pointes, or a history of long QT syndrome.
9. Medical history of difficulty swallowing, malabsorption or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product.
10. Anti-cancer treatment with radiation therapy, surgery, chemotherapy, targeted therapies (erlotinib, lapatinib, etc.), hormone therapy, or immunotherapy within 4 weeks (6 weeks for nitrosoureas or Mitomycin C) prior to trial entry, and ever use PARP inhibitor.
11. Participation in an investigational drug or device trial within 4 weeks prior to the trial entry.
12. Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
13. Recent venous thrombosis (including deep vein thrombosis or pulmonary embolism within 1 year of study).
14. History of upper gastrointestinal hemorrhage, peptic ulcer disease, or bleeding diathesis.
15. Subject is pregnant (positive serum beta human chorionic gonadotropin [β-HCG] test at screening) or is currently breast-feeding, their partner anticipates becoming pregnant/impregnating during the trial or within 6 months after receiving the last dose of trial treatment.
16. History of organ allograft, autologous stem cell transplantation, or allogeneic -
17. Concomitant disease or condition that could interfere with the conduct of the trial, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this trial.
18. Unwillingness or inability to comply with the trial protocol for any reason.
19. Legal incapacity or limited legal capacity.
20. Known drug abuse or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 4 weeks
  MTD will be defined as the maximum dose level at which no more than one 1 of 3 participants experience a dose-limiting toxicity (DLT) within the first 4 weeks of multiple dosing

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events | 24 months
Peak plasma concentration (Cmax) | 4 weeks
Area under the plasma concentration versus time curve (AUC） | 4 weeks
T1/2 (half-life) | 4 weeks
Clearance (CL) | 4 weeks
Volume of distribution at steady state (Vss) | 4 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Border Medical Oncology, Albury, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Linear, Melbourne

IPD SHARING:
Plan to Share IPD: No